CLINICAL TRIAL: NCT02728011
Title: A Double-Blind Randomized Pilot Trial Comparing Computerised Cognitive Exercises to Tetris in Adolescents With Attention-Deficit/Hyperactivity Disorder
Brief Title: Pilot Trial Comparing Computerised Cognitive Exercises to Tetris in Adolescents With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Syddanmark (Other)
Collaborators: Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Aida Bikic, psychologist, ph.d. candidate, Region Syddanmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7/6/2010
Record Dates: First submitted 2016-03-24; First posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Attention Deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Scientific Brain Training (SBT)
  Interventions: Other: Scientific Brain Training (SBT)
- Controle (Placebo Comparator): Tetris
  Interventions: Other: Tetris

INTERVENTIONS:
Other: Scientific Brain Training (SBT) — Cognitive training
  Arms: Intervention
Other: Tetris
  Arms: Controle

SUMMARY:
The purpose of this study was to examine the feasibility and efficacy of computerized cognitive exercises from Scientific Brain Training (SBT), compared to the computer game Tetris as an active placebo, in a pilot study of adolescents with Attention-deficit/hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
Objective: To examine the feasibility and efficacy of computerized cognitive exercises from Scientific Brain Training (SBT), compared to the computer game Tetris as an active placebo, in a pilot study of adolescents with Attention-deficit/hyperactivity disorder (ADHD).

Method: Eighteen adolescents with ADHD were randomized to treatment or control intervention for seven weeks. Outcome measures were cognitive test, symptom and motivation questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. a clinical diagnosis of hyperkinetic disorder (F90.0, corresponding to ADHD combined type) (WHO, 1993);
2. age between 14-17 years;
3. IQ > 80.

Exclusion Criteria:

1. pharmacological treatment other than methylphenidate, dexamphetamine and/or atomoxetine;
2. comorbid conduct disorder, autism spectrum disorders or major depression;
3. history of head trauma or verified neurological disease;
4. motor or perceptual disabilities which prevented the use of a computer;
5. medical illness that required treatment;
6. no access to a computer and internet at home.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Activity Perception Questionnaire | 7 weeks

SECONDARY OUTCOMES:
Attention Deficit/Hyperactivity Disorder-Rating Scale | 7 weeks
Cambridge Neuropsychological Test Automated Battery (CANTAB) Rapid Visual Information Processing (RVP)(A) | 7 weeks
CANTAB: Stockings of Cambridge (SOC) (problems solved in minimum moves) | 7 weeks
CANTAB: DMS Delayed Matching to Sample (DMS) | 7 weeks

OTHER OUTCOMES:
CANTAB: Spatial Span (SSP) | 7 weeks
CANTAB: Intra-Extra Dimensional Set Shift (IED) | 7 weeks
CANTAB: Spatial Working Memory (SWM) | 7 weeks
Cambridge Neuropsychological Test Automated Battery (CANTAB) Rapid Visual Information Probability of hit | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aida Bikic, MSc, Principal Investigator — Region Syddanmark
Locations (2):
- Denmark (2):
  - Child and Adolescent Mental Health Services Aabenraa, Aabenraa
  - Child and Adolescent Mental Health Services Augustenborg, Augustenborg

IPD SHARING:
Plan to Share IPD: Yes